CLINICAL TRIAL: NCT07222527
Title: A Randomized Trial of One vs. Two Transpapillary Cystic Duct Stents to Prevent Recurrent Symptomatic Gallbladder Disease in Non-Cholecystectomy Candidates
Brief Title: One vs. Two Stents for Gallbladder Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Eric J. Vargas Valls, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-011410; 95352001 (Other Grant/Funding Number: Mayo Clinic)
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Cholecystitis; Cholecystitis; Symptomatic Gallbladder Disease; Biliary Colic
Keywords: gallbladder disease; symptomatic gallbladder disease; Recurrent cholecystitis; biliary colic; cystic duct stent; transpapillary gallbladder stents; high surgical risk patient; nonsurgical management gallbladder disease; gallbladder decompression; acute cholecystitis in non-cholecystectomy candidate
MeSH Terms: conditions — Cholecystitis; Gallbladder Diseases | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ONE STENT ARM (Active Comparator): Participant assigned to this Arm will undergo ERCP and have one transpapillary duct stent placed for the treatment of symptomatic gallbladder disease
  Interventions: Procedure: ERCP with one stent placement
- TWO STENT ARM (Active Comparator): Participant assigned to this ARM will undergo ERCP and have two transpapillary duct stent placed for the treatment of symptomatic gallbladder disease.
  Interventions: Procedure: ERCP with two stent placement

INTERVENTIONS:
Procedure: ERCP with one stent placement — One transpapillary cystic duct stent will be placed into the gallbladder via ERCP
  Arms: ONE STENT ARM
Procedure: ERCP with two stent placement — Two transpapillary cystic duct stents will be placed into the gallbladder via ERCP
  Arms: TWO STENT ARM

SUMMARY:
This randomized trial will look at whether placing two cystic duct stents is more effective than one cystic duct stent in preventing recurrent gallbladder disease (cholecystitis, gallstone pancreatitis, or biliary colic) among patients who are not immediate surgical candidates for removal of their gallbladder.

The study will evaluate the safety profile, including rates of recurrent cholecystitis, biliary colic, and procedure-related complications, and technical success, defined as successful placement of stents into the gallbladder.

The main questions it aims to answer are:

1. Does placement of two transpapillary cystic duct stents reduce the risk of recurrent symptomatic gallbladder disease compared to one stent?
2. Is there a difference in procedure-related adverse events (post-ERCP pancreatitis, cholangitis, stent migration) between the two strategies?

Researchers will compare outcomes between patients randomized to one stent versus two stents to determine which approach provides better long-term gallbladder drainage and fewer recurrent events.

Participants will:

Be evaluated for eligibility and provide informed consent prior to undergoing an endoscopic retrograde cholangiopancreatography (ERCP), an endoscopy where a guidewire is placed into the bile duct from the small intestine.

They will then undergo ERCP with transpapillary cystic duct stent placement, randomized to one or two stents.

All participants will receive standard post-procedure care and follow-up assessments for recurrence, adverse events, and need for reintervention.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant females presenting with cholecystitis, biliary colic or gallstone pancreatitis.
2. Age 18-95.
3. Participants must be willing and able to provide informed consent
4. Referred for ERCP for management of 1) suspected choledocholithiasis 2) acute biliary pancreatitis and/or 3) acute cholangitis in whom cholecystectomy is expected to be delayed > 30 days or are deemed to not be surgical candidates for cholecystectomy.

Exclusion Criteria:

1. Inability to provide informed consent
2. History of surgically altered upper gastrointestinal anatomy (e.g. Roux-en-Y gastric bypass, Billroth I/II) precluding standard ERCP
3. History of primary sclerosing cholangitis
4. History of gallbladder cancer
5. History of cholecystectomy
6. Unsuccessful biliary cannulation during ERCP -

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2027-05-27 (Estimated); Study Completion 2028-05-27 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 6 months
  Defined as absence of recurrence of symptomatic gallbladder disease (cholecystitis, gallstone pancreatitis, or biliary colic) at 6 months post-procedure.

SECONDARY OUTCOMES:
Technical Success | 1 day
  Defined as the ability to place the allocated number of transpapillary double pigtail stents into the gallbladder.
Time to Recurrence | 6 months
  The amount of time (days) from the index procedure to when a recurrence occurs
Reintervention | 6 months
  The proportion of participants who receive another endoscopic procedure due to failure/adverse events related to the index procedure
Adverse Events | 6 months
  The type and severity of adverse events that occur related to the index procedure for stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Eric Vargas, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and outcomes will be shared after study approval of request from investigators by the study team
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after publication of results to 5 years after publication

REFERENCES:
- [Result] Storm AC, Vargas EJ, Chin JY, Chandrasekhara V, Abu Dayyeh BK, Levy MJ, Martin JA, Topazian MD, Andrews JC, Schiller HJ, Kamath PS, Petersen BT. Transpapillary gallbladder stent placement for long-term therapy of acute cholecystitis. Gastrointest Endosc. 2021 Oct;94(4):742-748.e1. doi: 10.1016/j.gie.2021.03.025. Epub 2021 Mar 30. PMID 33798540